CLINICAL TRIAL: NCT04510974
Title: Orthostatic Blood Pressure and Arterial Stiffness in Persons With SCI: The Effect of RAAS System
Brief Title: RAAS and Arterial Stiffness in SCI
Status: Completed | Type: Observational
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Kessler Foundation (Other); Seton Hall University (Other)
Responsible Party: Principal Investigator, Jill M. Wecht, Ed.D., Principal Investigator, James J. Peters Veterans Affairs Medical Center
Other Study IDs: WEC-18-025
Record Dates: First submitted 2020-08-10; First posted 2020-08-12 (Actual); Results first posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Arterial Stiffness; Renin Angiotensin Aldosterone System; Orthostatic Hypotension; Spinal Cord Injury; Hypotension
MeSH Terms: conditions — Hypotension, Orthostatic; Spinal Cord Injuries; Hypotension | interventions — Creb3l2 protein, rat

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cervical SCI: Ages between 21-70 years old Injured between C1-T1 Wheelchair dependent AIS classification of A, B or C Injury occurred more than 1 year ago
  Interventions: Other: Spinal Cord Injury
- Thoracic SCI: Ages between 21-70 Injured between T6-T12 Wheelchair dependent AIS classification of A, B or C Injury occurred more than 1 year ago
  Interventions: Other: Spinal Cord Injury
- Able-bodied Control: Ages between 21-70

INTERVENTIONS:
Other: Spinal Cord Injury — Spinal Cord Injury
  Groups: Cervical SCI; Thoracic SCI

SUMMARY:
The study is examining differences in central arterial stiffness, orthostatic changes in blood pressure, norepinephrine, and plasma renin in individuals with spinal cord injury compared with age-matched uninjured controls.

DETAILED DESCRIPTION:
The study is examining differences in central arterial stiffness, orthostatic changes in blood pressure, norepinephrine, and plasma renin in individuals with spinal cord injury compared with age-matched uninjured controls. Arterial stiffness and blood pressure will be collected in the laying down position. A blood sample of norepinephrine and plasma renin will also be collected. The participant will tilt to 30, 45 and 60 degrees for 10 minutes at each angel. Blood pressure and heart rate will be monitored at each angle. Another blood sample of renin and norepinephrine will be collected at the end of 10 minutes at 60 degrees.

ELIGIBILITY:
Inclusion Criteria:

* SCI participants:
* injured between C1-T1 and T6-T12
* wheelchair dependent
* AIS classification A, B or C
* Injured occurred more than 1 year ago

Exclusion Criteria:

* currently have an illness or infection
* current smoker of at least 1 year
* controlled or uncontrolled hypertension or diabetes mellitus
* Neurological condition other than SCI (Alzheimer's disease, dementia, stroke, multiple sclerosis, Parkinson's disease)
* cardiovascular disease (coronary heart disease, congestive heart failure, peripheral artery disease)

Ages: 21 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Outpatient individuals with SCI, flyers in town
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2018-06-30 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- James J Peters VAMC, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cervical SCI | Thoracic SCI | Able-bodied Control
Started | 11 | 11 | 11
Completed | 11 | 11 | 11
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervical SCI | Thoracic SCI | Able-bodied Control | Total
Number analyzed (Participants) | 11 | 11 | 11 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 11 | 33
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (13) | 43 (11) | 45 (13) | 44 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 2 | 7
  Male | 8 | 9 | 9 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 3
  Not Hispanic or Latino | 9 | 11 | 10 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 11 | 33

OUTCOME MEASURES:

1. Primary Outcome: Pulse Wave Velocity (m/s)
Description: Determine average pulse wave velocity among the three groups.
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Cervical SCI | Thoracic SCI | Able-bodied Control
Number analyzed (Participants) | 11 | 11 | 11
m/s | 8.81 (1.91) | 7.36 (1.58) | 5.53 (0.95)

2. Secondary Outcome: Systolic Blood Pressure (mmHg)
Description: Determine differences in blood pressure among groups
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Cervical SCI | Thoracic SCI | Able-bodied Control
Number analyzed (Participants) | 11 | 11 | 11
mmHg | 95 (20) | 125 (14) | 128 (27)

3. Secondary Outcome: Plasma Renin (pg/ml)
Description: Determine differences in plasma renin among the groups
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Cervical SCI | Thoracic SCI | Able-bodied Control
Number analyzed (Participants) | 11 | 11 | 11
pg/mL | 24.9 (13.9) | 21.9 (18) | 16.0 (7.4)

4. Secondary Outcome: Norepinephrine (pg/ml)
Description: Determine differences in plasma norepinephrine among the groups.
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Cervical SCI | Thoracic SCI | Able-bodied Control
Number analyzed (Participants) | 11 | 11 | 11
pg/mL | 176.0 (90.0) | 515.6 (162.3) | 371.8 (118.3)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Cervical SCI | Thoracic SCI | Able-bodied Control
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-06): https://cdn.clinicaltrials.gov/large-docs/74/NCT04510974/Prot_SAP_000.pdf